CLINICAL TRIAL: NCT03097341
Title: A Phase 1, Single Ascending Dose, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Xisomab 3G3 in Healthy Adult Subjects
Brief Title: Safety and Tolerability Study of Xisomab 3G3 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aronora, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3G3-15-01
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- xisomab 3G3- Dose 1 (Experimental): Participants will receive a single intravenous dose of 0.1 mg/kg xisomab 3G3.
  Interventions: Drug: xisomab 3G3- Dose 1
- xisomab 3G3- Dose 2 (Experimental): Participants will receive a single intravenous dose of 0.5 mg/kg xisomab 3G3.
  Interventions: Drug: xisomab 3G3-Dose 2
- xisomab 3G3- Dose 3 (Experimental): Participants will receive a single intravenous dose of 2.0 mg/kg xisomab 3G3.
  Interventions: Drug: xisomab 3G3-Dose 3
- xisomab 3G3- Dose 4 (Experimental): Participants will receive a single intravenous dose of 5.0 mg/kg xisomab 3G3.
  Interventions: Drug: xisomab 3G3- Dose 4
- Placebo (Placebo Comparator): Participants will receive a single intravenous dose of placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: xisomab 3G3- Dose 1 — Participants will receive a single intravenous dose of 0.1 mg/kg xisomab 3G3.
  Other Names: AB023- Dose 1
  Arms: xisomab 3G3- Dose 1
Drug: xisomab 3G3-Dose 2 — Participants will receive a single intravenous dose of 0.5 mg/kg xisomab 3G3.
  Other Names: AB023- Dose 2
  Arms: xisomab 3G3- Dose 2
Drug: xisomab 3G3-Dose 3 — Participants will receive a single intravenous dose of 2.0 mg/kg xisomab 3G3.
  Other Names: AB023- Dose 3
  Arms: xisomab 3G3- Dose 3
Drug: xisomab 3G3- Dose 4 — Participants will receive a single intravenous dose of 5.0 mg/kg xisomab 3G3.
  Other Names: AB023- Dose 4
  Arms: xisomab 3G3- Dose 4
Other: Placebo — Participants will receive a single intravenous dose of placebo.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of xisomab 3G3 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or female (non-childbearing potential only), 18 to 48 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine containing products for at least 3 months prior to dosing and throughout the study.
3. Body mass index (BMI) ≥ 19 and ≤ 29.0 (kg/m2) and weight between 50 and 125 kg (inclusive) at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), lactate dehydrogenase (LDH), blood urea nitrogen (BUN), creatinine must be between the lower limit of normal (LLN; or up to 15% below LLN as not indicative of hepatic or renal disease in healthy subjects) and the upper limit of normal, inclusive, at screening and check-in.
6. aPTT, PT/INR, and platelets, must be within the limits of normal, inclusive, at screening and check-in.
7. Bleeding time must be between 2 to 8 minutes, inclusive, at check-in.
8. For a female of non childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to dosing:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to dosing and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.
9. A non vasectomized male subject whose sexual partner is sterile or was advised to use one of the following during the course of the study (or prior to study as specified) and for 90 days following dosing:

   * Abstain from sexual intercourse;
   * An intrauterine device with spermicide;
   * A physical barrier method (e.g., male or female condom, contraceptive sponge, diaphragm, cervical cap) with spermicide;
   * An intravaginal system (e.g., NuvaRing®) for at least 3 months prior to dosing;
   * An oral, implantable, transdermal, or injectable hormonal contraceptive for at least 3 months prior to dosing.

   No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to dosing. A male who has been vasectomized less than 4 months prior to dosing must follow the same restrictions as a non vasectomized male.
10. If male, must agree to not donate sperm from dosing until 90 days after dosing.
11. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of drug abuse within the last 2 years prior to dosing.
5. History of alcoholism within the last 2 years prior to dosing or a current history of imbibing 3 or more units of alcohol per day (1 unit is equivalent to 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol).
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drug, any ingredients of the study drug, or related compounds.
7. History of a clinically significant allergy of any kind including a history of allergic or hypersensitivity reactions to any drugs.
8. History or presence of:

   * Bleeding disorder(s) and/or at risk of bleeding, including relevant familial history;
   * Clinically significant anemia, in the opinion of the PI or designee;
   * Thromboembolic disease;
   * Bleeding in the gastrointestinal tract or central nervous system.
9. Allergy to rodents.
10. Had a minor surgery or major physical injury less than 4 weeks or major surgery less than 12 weeks prior to screening.
11. Was hospitalized within 2 months of dosing, unless deemed acceptable by the PI or designee.
12. Female subjects of childbearing potential.
13. Female subjects who are pregnant or lactating.
14. Positive urine drug or alcohol results at screening or check in.
15. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
16. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
17. Seated heart rate is lower than 40 bpm or higher than 100 bpm at screening.
18. QTcF interval is >450 msec (males) or >460 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
19. Hemoglobin value of less than 11.5 g/dL for females and 13.0 g/dL for males, at screening or check-in.
20. Unable to refrain from or anticipates the use of:

    * Any prescription medications, non-prescription medications, herbal remedies, or vitamin supplements beginning approximately 14 days prior to dosing and throughout the study. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study and will be documented.
    * Any anticoagulants (i.e., warfarin, Low Molecular Weight Heparin), coagulants, anti-platelet (e.g., clopidogrel), nonsteroidal anti-inflammatory drugs and/or acetylsalicylic acid beginning approximately 28 days prior to dosing and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of pharmacokinetic/pharmacodynamic interaction with study drug.
    * Any investigational drugs or biologics beginning approximately 30 days prior to dosing and throughout the study.
    * Any biologics developed from chinese hamster ovary cell cultures in their life time.
21. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 28 days prior to dosing and throughout the study.
22. Donation of blood or significant blood loss within 56 days prior to dosing.
23. Plasma donation within 7 days prior to dosing.
24. Strenuous exercise/physical activity which could cause muscle aches or injury, including contact sports at any time from 72 hours before dosing until completion of the study.
25. Participation in another clinical study within 30 days prior to dosing. The 30 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study.
26. Presence of any scars, or tattoos which may obscure the injection site, as deemed by PI or designee.
27. Any condition or circumstance, in the opinion of the PI or designee, which may make the subject unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the subject's safety.

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Lorentz CU, Verbout NG, Wallisch M, Hagen MW, Shatzel JJ, Olson SR, Puy C, Hinds MT, McCarty OJT, Gailani D, Gruber A, Tucker EI. Contact Activation Inhibitor and Factor XI Antibody, AB023, Produces Safe, Dose-Dependent Anticoagulation in a Phase 1 First-In-Human Trial. Arterioscler Thromb Vasc Biol. 2019 Apr;39(4):799-809. doi: 10.1161/ATVBAHA.118.312328. PMID 30700130

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 105 participants were screened for the study, of which 84 did not meet eligibility criteria or declined to participate. The remaining 21 participants were randomized into the study, with each dose level occurring in sequential order.
Groups:
- Xisomab 3G3- Dose 1: Participants received a single intravenous dose of 0.1 mg/kg xisomab 3G3.
- Xisomab 3G3- Dose 2: Participants received a single intravenous dose of 0.5 mg/kg xisomab 3G3.
- Xisomab 3G3- Dose 3: Participants received a single intravenous dose of 2.0 mg/kg xisomab 3G3.
- Xisomab 3G3- Dose 4: Participants received a single intravenous dose of 5.0 mg/kg xisomab 3G3.
- Placebo: Participants received a single intravenous dose of placebo.
Period: Overall Study
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Started | 4 | 4 | 4 | 4 | 5
Completed | 4 | 4 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5 | 21
Age, Continuous [Mean (Full Range); unit: years] | 42.3 [37 to 47] | 33.0 [25 to 46] | 32.0 [22 to 42] | 42.0 [40 to 45] | 32.2 [25 to 42] | 36.1 [22 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 1 | 2 | 9
  Male | 1 | 2 | 3 | 3 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 3 | 4 | 17
  Not Hispanic or Latino | 0 | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 4 | 3 | 4 | 3 | 5 | 19
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 5 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Treatment-related Adverse Events (TEAEs) Will be Summarized Using Frequency Counts.
Description: TEAEs will be determined by physical examination that will include assessment of skin, head, ears, eyes, nose, throat, respiratory system, cardiovascular system, gastrointestinal system, neurological condition, blood and lymphatic systems, and the musculoskeletal system.
Time Frame: From Subject Check-In through Follow up. Follow up was performed 7 days after Day 29. If the aPTT was not +/- 10% baseline or within normal range, subject was monitored weekly until baseline reached and follow up then occured 7 days after.
Population: Subjects who received any dose of study drug or placebo were included in the as-treated population and subjects were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 1 | 3 | 1 | 2 | 3

2. Primary Outcome: The Number of Subjects With Abnormal Vital Signs That Are Related to Treatment Will be Summarized Using Frequency Counts..
Description: Vital sign measurements (body temperature, respiratory rate, blood pressure, and heart rate)
Time Frame: as for outcome 1
Population: Subjects who had received any dose of study drug were included in the as-treated population and subjects were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: The Number of Subjects With Abnormal Electrocardiogram That is Related to Treatment Will be Summarized Using Frequency Counts..
Description: 12-lead electrocardiogram measurement
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: The Number of Subjects With Abnormal Injection Site Reaction That Are Related to Treatment Will be Summarized Using Frequency Counts..
Description: Injection site reaction (pain, tenderness, erythema/ redness, and induration/ swelling)
Time Frame: From Study Day 1 through Follow up. Follow up was performed 7 days after Day 29. If the aPTT was not +/- 10% baseline or within normal range, subject was monitored weekly until baseline reached and follow up then occured 7 days after.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 1 | 0 | 0 | 0

5. Primary Outcome: The Number of Subjects With Abnormal Laboratory Values and/ or Adverse Events That Are Related to Treatment Will be Summarized Using Frequency Counts..
Description: Clinical laboratory tests include serum chemistry, hematology, coagulation parameters (aPTT, PT, and bleeding time), and urinalysis
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: The Number of Subjects That Develop Treatment-related Immunogenicity Will be Summarized Using Frequency Counts.
Description: Immunogenicity measured by the presence of plasma anti-drug antibodies
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
Participants
  Pre-dose (baseline) | 0 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0 | 0
  Day 29 or follow up | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: The Maximum Plasma Concentration (Cmax) of Xisomab 3G3 After a Single Injection Will be Measured in Each Subject.
Description: Maximum plasma concentration of xisomab 3G3 was estimated based on plasma xisomab 3G3 concentrations. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: Pre-dose (0.5h prior to dose), 0.083, 0.25, 0.5, 1,3,8,24,72,120, 168, 216, 336, 504, 672h after dosing as well as follow up (7 days after aPTT returned back to baseline).
Population: All subjects who were enrolled in, received the active treatment, completed the study, and had an evaluable PK profile were included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 3 | 4 | 4 | 4
nanograms/milliliter | 122.7 (23.3) | 11210 (9.1) | 42510 (12.3) | 127200 (2.6)

8. Secondary Outcome: The Time to Reach Maximum Plasma Concentrations of Xisomab 3G3 (Tmax) After a Single Injection Will be Measured in Each Subject.
Description: The time to reach maximum plasma concentrations of xisomab 3G3 after a single injection was estimated based on plasma xisomab 3G3 concentrations. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 3 | 4 | 4 | 4
hours | 0.084 [0.08 to 0.09] | 0.649 [0.26 to 3.02] | 0.088 [0.08 to 0.25] | 0.387 [0.26 to 3.00]

9. Secondary Outcome: The Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Non-zero Concentration (AUC0-t), as Calculated by the Linear Trapezoidal Method, After a Single Injection of Xisomab 3G3 Will be Calculated for Each Subject.
Description: The area under the plasma concentration-time curve from time 0 to the last measurable non-zero concentration was estimated based on plasma xisomab 3G3 concentrations. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanograms*hour/milliliter
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 3 | 4 | 4 | 4
nanograms*hour/milliliter | 57.0 (46.5) | 361800 (21.9) | 5540000 (23.9) | 28120000 (11.8)

10. Secondary Outcome: The Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) After a Single Injection of Xisomab 3G3 Will be Calculated for Each Subject.
Description: The area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) is calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 1 | 4 | 4 | 4
nanogram*hour/milliliter | 184.7 | 363700 (21.8) | 5550000 (24.0) | 28140000 (11.8)

11. Secondary Outcome: The Percent of AUC0-inf Extrapolated (AUC%Extrap) After a Single Injection of Xisomab 3G3 Will be Calculated for Each Subject.
Description: The percent of AUC0-inf extrapolated (AUC%extrap) is calculated by (1-AUC0-t/AUC0-inf)*100. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of AUC0-inf
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 1 | 4 | 4 | 4
percentage of AUC0-inf | 57.3 | 0.53 (0.18) | 0.18 (0.07) | 0.07 (0.04)

12. Secondary Outcome: The Apparent First Order Terminal Elimination Rate Constant (Kel) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Subject.
Description: The apparent first order terminal elimination rate constant will be calculated from a semi-log plot of the plasma concentration versus time curve. The parameter will be calculated by linear least squares regression analysis using the maximum number of points in the terminal log linear phase (e.g., three or more non zero plasma concentrations). Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 1 | 4 | 4 | 4
1/hour | 0.522 | 0.042 (0.0042) | 0.011 (0.0009) | 0.006 (0.0018)

13. Secondary Outcome: The Apparent First Order Terminal Elimination Half-life (T1/2) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Subject.
Description: The apparent first order terminal elimination half-life will be calculated as 0.693/Kel. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 1 | 4 | 4 | 4
hours | 1.33 | 16.64 (1.56) | 60.63 (4.45) | 121.49 (40.69)

14. Secondary Outcome: The Apparent Total Plasma Clearance (CL) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Subject.
Description: The apparent total plasma clearance will be calculated as [Dose/AUC0-inf]. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 1 | 4 | 4 | 4
Liters/hour | 37.46 | 0.094 (0.018) | 0.026 (0.003) | 0.014 (0.003)

15. Secondary Outcome: The Total Apparent Volume of Distribution (Vss) of Xisomab 3G3 After a Single Intravenous Injection Will be Calculated for Each Subject.
Description: The total apparent volume of distribution (Vss) will be calculated as the mean residence time x clearance. Non-compartmental PK data analysis was performed to estimate the plasma PK parameters of xisomab 3G3.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4
Number analyzed (Participants) | 1 | 4 | 4 | 4
Liters | 69.11 | 2.52 (0.59) | 3.72 (0.42) | 4.31 (0.75)

16. Secondary Outcome: The Effect of a Single Intravenous Dose of Xisomab 3G3 on the Activated Partial Thromboplastin Time (aPTT) in Healthy Adult Subjects Will be Measured.
Description: Activated partial thromboplastin time (aPTT) will be used as a surrogate pharmacodynamic marker.
Time Frame: Pre-dose (0.5h prior to dose), 1, 24,72, 168, 336, 504, 672h after dosing as well as follow up (7 days after day 29 or after aPTT returned back to baseline)..
Population: All subjects who had received any dose of study drug were included in the as-treated population and subjects were analyzed according to treatment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 5
seconds
  pre-dose | 27.0 (1.8) | 26.5 (1.3) | 26.3 (2.6) | 27.5 (1.7) | 29.4 (1.7)
  Day 1, Hour 1 | 32.8 (3.8) | 48.3 (0.5) | 53.3 (5.7) | 57.3 (7.8) | 29.4 (1.7)
  Day 2 | 29.0 (2.3) | 50.5 (5.8) | 52.5 (4.8) | 55.8 (6.9) | 28.8 (2.0)
  Day 4 | 28.3 (2.6) | 48.8 (6.5) | 49.8 (3.9) | 52.3 (5.6) | 27.3 (2.1)
  Day 8 | 27.3 (2.1) | 30.5 (3.9) | 47.3 (2.2) | 49.8 (5.3) | 28.6 (1.1)
  Day 15 | 26.8 (2.1) | 27.5 (2.1) | 47.0 (2.9) | 48.0 (6.5) | 29.0 (1.2)
  Day 22 | 26.5 (2.4) | 27.5 (2.6) | 39.5 (6.6) | 48.3 (6.3) | 28.8 (0.8)
  Day 29 | 27.0 (2.3) | 27.5 (2.1) | 30.3 (2.9) | 47.3 (5.0) | 29.2 (1.3)
  Follow Up | 26.8 (1.5) | 27.3 (1.7) | 28.3 (1.5) | 28.0 (2.2) | 29.2 (1.3)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from subject check-in through follow-up. Follow-up was performed 7 days after day 29. Subjects for whom aPTT did not reach +/- 10% of baseline or within normal range by Study Day 29 returned every 7 days until aPTT reached within +/- 10% of baseline or within normal range and the follow up visit was conducted 7 days after it was reached.
Arm/Group | Xisomab 3G3- Dose 1 | Xisomab 3G3- Dose 2 | Xisomab 3G3- Dose 3 | Xisomab 3G3- Dose 4 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/4 | 3/4 | 1/4 | 2/4 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xisomab 3G3- Dose 1 (N=4) | Xisomab 3G3- Dose 2 (N=4) | Xisomab 3G3- Dose 3 (N=4) | Xisomab 3G3- Dose 4 (N=4) | Placebo (N=5)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site ecchymosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — administration site condition
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — administration site condition
Upper respiritory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oralpharangeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Aronora shall retain title to and the right to publish all documentation, records, raw data, specimens or other work product generated in connection with this study. Such publications shall not be made by the PI or Celerion without the prior written consent of Aronora.

DOCUMENTS (2):
  • Study Protocol (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03097341/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT03097341/SAP_001.pdf